CLINICAL TRIAL: NCT04259736
Title: A Prospective Cohort Study of Molecular Mechanism of Lower Respiratory Tract Microbes in Patients With Acute Obstructive Pulmonary Disease (AECOPD) by Regulating the Transcriptional Balance of NF-κB and PPARγ in Alveolar Macrophages
Brief Title: Prospective Cohort Study of Molecular Mechanism of Lower Respiratory Tract Microbes in Patients With AECOPD
Acronym: REASON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Shengqing Li, Chief Physician,Professor, Huashan Hospital
Other Study IDs: KY2018-362
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Microbiome
Keywords: Lower Respiratory Tract; Microbes; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Specimens include blood specimens and alveolar lavage fluid, used to detect blood routine, peripheral blood inflammatory factors (IL-8, TNF-α, IL-17), alveolar tube lavage microorganisms, and alveolar lavage fluid inflammatory factors (NF- κB, PPARγ, MMP-12, TIMP-4).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
How to reduce the rapid decline of lung function in patients with AECOPD is a clinically urgent problem to be solved. Studies have suggested that there is a bacterial flora imbalance in the lower respiratory tract of COPD patients. To explore the relationship between microbiology and host immunity is a hot topic in the field of COPD. The investigators use NGS (next generation sequencing) technology to fully explore the specific molecular mechanism of the lower respiratory tract microbiome in patients with COPD by regulating the transcriptional activities of NF-κB and PPARγ in alveolar macrophages, resulting in pulmonary parenchymal remodeling and decreased lung function. In this study, a prospective cohort study will be used to evaluate the effect of the lower respiratory tract microbiome on lung tissue (alveolar space and pulmonary vascular) remodeling and pulmonary function decline in patients with AECOPD.

DETAILED DESCRIPTION:
This study will be based on a prospective cohort design in patients with COPD who are eligible for the study. Fifty patients who met the criteria for inclusion and exclusion of COPD exacerbations and signed informed consent will participate in the study. The purpose of this study is to evaluate the effect of the lower respiratory tract microbiome on lung tissue remodeling, decreased lung function, and clinical symptoms in patients with AECOPD.

Baseline screening includes demographic data, medical history, combined medication records, symptoms, signs, symptom scores, number of acute exacerbations, blood cells and inflammatory factors, electrocardiogram, lung function, alveolar lavage fluid microbe NGS, and safety observation indicators.

Patients will be followed up every 3 months for a period of 1 year. The primary and secondary endpoints are as follows.

Primary endpoint： Changes in FEV1 (forced expiratory volume in the first second) within 1 year of follow-up

Secondary endpoint： Changes in CAT, CCQ, mMRC scores during 1 year of follow-up Changes in lung function during 1 year of follow-up: FEV1 / FVC Changes in blood routine, IgE, and eosinophil count within 1 year of follow-up Number of hospital admissions due to acute exacerbation during 1 year of follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of acute exacerbation of chronic obstructive pulmonary disease (AECOPD) according to the GOLD2018 guidelines (patients with FEV1pred> 30% and no concurrent respiratory failure);
2. Age ≥18, ≤80 years, regardless of gender;
3. No antibiotics have been used after this acute exacerbation;
4. Treatment according to GOLD guidelines;
5. Those with the following bronchoscopy indications:

   1. Collect lower respiratory tract secretions for bacteriological examination;
   2. Chest radiographs have invasive lesions of unknown origin;
   3. bronchoalveolar lavage, bronchial administration and suction treatment;
   4. unexplained hemoptysis or chronic irritating cough;
   5. Bronchial obstructions such as localized wheezing, localized emphysema, obstructive pneumonia, or any atelectasis;
   6. Suspected of trachea and bronchial tumors;
   7. paralysis of the recurrent laryngeal or phrenic nerve of unknown cause;
   8. Cancer cells or Mycobacterium tuberculosis are found in sputum and no lesions are found on chest radiograph;
   9. Suspected of bronchial foreign bodies or stones;
   10. diffuse lesions of the lungs or masses around the lungs that require lung biopsy, brushing, or lavage for cytology or bacteriological examination to confirm the diagnosis;
   11. Patients who have a long-term indwelling cannula after tracheotomy and know whether the trachea is damaged or necrotic;
   12. hilar swollen, unexplained lung mass;
   13. Select lipiodol or iodine radiography of a lung lobe or segment.
6. Voluntary signed informed consent.

Exclusion Criteria:

1. active phase of tuberculosis;
2. Patients with malignant tumor disease;
3. patients with rheumatic diseases;
4. Patients with contraindications to bronchoscopy;
5. patients with mental illness;
6. Exclude those with severe medical diseases: such as heart, liver, and kidney dysfunction or coagulation dysfunction; uncontrolled hypertension, hyperglycemia or arrhythmia;
7. pregnancy and lactation;
8. Patients who participated in other clinical trials in the past 3 months;
9. Staff members and their families in this research institution.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty patients who met the criteria for inclusion and exclusion of COPD exacerbations and signed informed consent will participate in the study. Patients will be followed up every 3 months for a period of 1 year.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 12 months
  Forced expiratory volume in the first second

SECONDARY OUTCOMES:
CAT scores | 12 months
  COPD Assessment Test score; Score: 0-10, Low impact; Score: 10-20, Moderate impact; Score 20-30, High impact; Score 30-40, Very high impact.
mMRC scores | 12 months
  The modified British Medical ResearchCouncil (mMRC) questionnaire total score ranges from 0 to 4, with higher grades indicating more severe breathlessness.
other lung function parameters | 12 months
  FEV1/ FVC
Incidence of COPD exacerbation | 12 months
  Number of Incidence of COPD exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital,Fudan university, Shanghai, Shanghai Municipality, China